CLINICAL TRIAL: NCT06754917
Title: Feasibility Testing of the "Face-Forward-Web" Program for Chronic Orofacial Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Jonathan Greenberg, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024P003501; 1R21DE033502-01A1 (NIH)
Record Dates: First submitted 2024-12-23; First posted 2025-01-01 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Orofacial Pain; Facial Pain
Keywords: Chronic orofacial pain; Facial Pain; Mindfulness; web-based delivery
MeSH Terms: conditions — Facial Pain

STUDY DESIGN:
Intervention Model Description: NIH Stage Model for Behavioral Intervention Development
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Face-Forward-Web (Experimental): A 5-session web-based mind-body pain management intervention focused on decreasing pain and disability (physical and emotional) among adult patients with chronic orofacial pain.
  Interventions: Behavioral: Face-Forward-Web

INTERVENTIONS:
Behavioral: Face-Forward-Web — This is a self-administered web-based mind-body intervention that consists of 5 30-minute video sessions disseminating tailored relaxation, mindfulness, and cognitive-behavioral skills for COP. Ultimately, the Face-Forward-Web program aims to increase patients' physical and emotional functioning and decrease pain intensity and maladaptive coping behaviors.

SUMMARY:
The goal of this study is to conduct a feasibility open pilot study (N=Up to 20) with exit interviews to assess the feasibility, acceptability, and credibility of the study protocol and Face-Forward-Web; a web-based mind-body intervention for adult patients with COP.

Deliverables: [1] Adapt and refine open pilot protocol, patient recruitment, and other study materials. [2] Assess the feasibility, acceptability, and credibility of Face-Forward-Web and optimize the intervention methodology in preparation for a future efficacy study.

This research leverages mixed methods information to evaluate the feasibility, acceptability, and credibility of Face-Forward-Web and optimize the intervention and study methodology in preparation for the subsequent pilot study and again later, for a pilot feasibility randomized control trial (RCT).

DETAILED DESCRIPTION:
Aim: Conduct a feasibility open pilot study (N=Up to 20) with exit interviews of Face-Forward-Web among adults with various chronic orofacial pain (COP). The ultimate goal of this research is to assess the feasibility, credibility, and acceptability of Face-Forward-Web and optimize the program and study methodology in preparation for a pilot feasibility randomized control trial (RCT).

Face-Forward-Web, adapted from GetActive (a mind-body program for patients with chronic musculoskeletal pain), is a mind-body program for COP and consists of 5 on-demand sessions over a web platform, each being approximately 30 minutes long. The program will teach relaxation (deep breething), mindfulness, and cognitive-behavioral skills to reduce pain and improve emotional welbeing in patients with COP. At the conclusion of each session, an interactive quiz covering the session's content is given to foster a stronger, and more long term, understanding of the material. Throughout the program, encouragements to practice and track the use of Face-Forward-Web skills are disseminated outside and/or between sessions through a variety of means (e.g, text, phone call, email), depending on individual preferenes. Home practice materials include Web-based audio and video clips (e.g., 5 min mindfulness of pain for COP) but, engagement in self-guided skill practice is also permitted.

Following program completion, there will be a one-time 15-30 minute exit interview to elicit subject perceptions of Face-Forward-Web and any recommendations to improve intervention quality. This information will be used to further adapt and optimize Face-Forward-Web prior to future efficacy testing.

Assessments: Baseline (0 weeks), post-test (5 weeks), and 3-month follow-up (17 weeks) survey assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18
2. English fluency and literacy
3. Nonmalignant chronic (>3 months) orofacial pain
4. Ability and willingness to participate in the Face-Forward web-platform intervention
5. Free of concurrent psychotropic medication 2 week prior to participation OR stable psychotropic medication dose and type for ≥ 6 weeks
6. Pain score ≥4/10 on the Numerical Rating Scale
7. Owns (or has easy access to) a device with internet access

Exclusion Criteria:

1. Practice of mindfulness > 45 minutes/week in the past 3 months
2. Participation in mind-body or cognitive-behavioral therapy in the past 3 months
3. Severe untreated mental health disorder (e.g., psychosis)
4. Active suicidal ideation with plan or intent
5. Pregnancy

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Who Scored Above the Midpoint on Each Subscale of the Credibility and Expectancy Questionnaire | Baseline (0 Weeks)
  Assessed using the Credibility and Expectancy Questionnaire which asks the participant to indicate how much they believe, right now, that the intervention they will receive will help manage their COP and related worry. Possible scores range from 3 to 27 for both the credibility and the expectancy subscales. Higher scores represent higher credibility and expectancy.
Proportion of Participants Who Scored Above the Midpoint on the Client Satisfaction Scale | Post-Test (5 Weeks)
  Measured using the Client Satisfaction Scale which assess participants' satisfaction with participation in the study. The score range is 0-12. Higher scores indicate greater satisfaction.
Feasibility of recruitment | Baseline (0 Weeks)
  The percent of eligible patients approached that agree to participate.
The User Experience Scale to assess participants' satisfaction with (acceptability of) web-based delivery | Post-Test (5 Weeks)
  This measure will assess how well patients like the Wed-based program content and delivery. Total raw scores range from 22 to 110 with higher scores indicating greater satisfaction with the platform.
Rate at which program was accepted, measured by number of completed program sessions | Post-Test (5 Weeks)
  The proportion of participants who complete > or = 3 of 5 sessions.
Adherence to homework | Collected during intervention, an average of 5 weeks
  Rate of participant's completion of homework assigned (practicing at least 1 program skill, 3 days/week on average) throughout the study
Feasibility of Assessments at Baseline | Baseline (0 Weeks)
  Rate of participant's completion of self-report measures, with no measures missing.
Feasibility of Assessments at Post-Test | Post-Test (5 Weeks)
  Rate of participant's completion of self-report measures, with no measures missing.
Feasibility of Assessments at Follow-Up | Follow-Up (17 Weeks)
  Rate of participant's completion of self-report measures, with no measures missing.
Adverse Events | Collected during intervention, an average of 5 weeks
  Any self-reported or observed negative events related to participation

OTHER OUTCOMES:
Graded Chronic Pain Scale (GCPS) | Baseline (0 Weeks), Post-Test (5 Weeks), Follow-Up (17 Weeks)
  A 7-item scale measuring pain severity and pain-related activity limitations. The time frame of reference will be the past week, consistent with prior work. This measure includes a pain intensity subscale and a pain interference subscale. Each subscale has a range of 0 to 100 with higher scores suggesting worse outcomes.
Applied Mindfulness Process Scale (AMPS) | Baseline (0 Weeks), Post-Test (5 Weeks), Follow-Up (17 Weeks)
  A 15-item questionnaire representing three domains of applied mindfulness processes (decentering, positive emotion regulation, negative emotion regulation) measuring the application of mindfulness practices in daily life among persons participating in mindfulness-based interventions. Total scores range from 0-60 with higher scores suggesting greater application of the use of mindfulness skills in daily life coinciding with mindfulness practice.
Cognitive And Affective Mindfulness Scale-Revised (CAMS-R) | Baseline (0 Weeks), Post-Test (5 Weeks), Follow-Up (17 Weeks)
  Rate of a participant's broad conceptualization of mindfulness, items range from 1-4 and scores range from 12-48, with higher values reflecting higher levels of mindfulness.
Tampa Scale for Kinesiophobia for Temporomandibular Disorders (TSK-TMD) | Baseline (0 Weeks), Post-Test (5 Weeks), Follow-Up (17 Weeks)
  An 18-item scale assessing fear of pain due to movement, adapted to heterogeneous facial pain (i.e., expanding references from "jaw" to "jaw or face". Scores for each item range from 1 to 4, with greater scores reflecting more severe kinesiophobia.
Pain Catastrophizing Scale (PCS) | Baseline (0 Weeks), Post-Test (5 Weeks), Follow-Up (17 Weeks)
  A 13-item questionnaire assessing one's tendency to focus on pain-related thoughts and feel helpless and hopeless due to pain on a scale of 0 to 4. Total scores range from 0 to 25 and higher scores indicate higher pain catastrophizing (worse outcomes).
Generalized Anxiety Disorder Scale (GAD-7) | Baseline (0 Weeks), Post-Test (5 Weeks), Follow-Up (17 Weeks)
  7-item questionnaire measuring symptoms of anxiety within the past 2 weeks on a scale of 0 to 3. Total scores range from 0 to 21 and higher scores indicate more symptoms of anxiety.
Patient Health Questionnaire - Depression (PHQ-9) | Baseline (0 Weeks), Post-Test (5 Weeks), Follow-Up (17 Weeks)
  A 9-item measure assessing symptoms of depression on a scale of 0 to 3. Higher scores equate to more depression symptoms.
Numerical Rating Scale (NRS) | Baseline (0 Weeks), Post-Test (5 Weeks), Follow-Up (17 Weeks)
  Self-reported pain score on a Likert scale with 0 being no pain and 10 being worst possible pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
The digital qualitative and quantitative data associated with this study will be shared by depositing these data in the Vivli database. Vivli is one of the recommended databases for similar NIH-funded chronic pain studies (including as part of the NIH HEAL initiative), with data types similar to the current study. Documentation and de-identified data will be deposited, including qualitative and quantitative data as well as demographics. Submitted data will conform with relevant data and terminology standards.

REFERENCES:
- [Derived] Lovette BC, Bakhshaie J, Kulich R, Shaefer JR, Cheng HT, He S, Vranceanu AM, Greenberg J. Development of a Novel Web-Based Intervention Targeting Pain-Related Outcomes in Individuals With Chronic Orofacial Pain: Protocol for a Mixed Methods Study. JMIR Res Protoc. 2025 Aug 20;14:e71839. doi: 10.2196/71839. PMID 40835226